CLINICAL TRIAL: NCT00346229
Title: A Phase I, Dose Escalation and Pharmacokinetics Study of Temperature Sensitive Liposome Encapsulated Doxorubicin (ThermoDox™) and Hyperthermia in Patients With Local-Regionally Recurrent Breast Cancer
Brief Title: Temperature-Sensitive Liposomal Doxorubicin and Hyperthermia in Treating Women With Locally Recurrent Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00014340; DUMC-6883-06-2R1; DUMC-06068; CDR0000482411 (Other: Secondary ID)
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer
Keywords: stage III B breast cancer; stage III C breast cancer; stage IV breast cancer; inflammatory breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Filgrastim; pegfilgrastim; Diathermy

ARMS (1):
- Thermodox (Experimental): ThermoDox20-40mg/m2 every 21-35 days followed by Chest Wall Hyperthermia
  Interventions: Biological: filgrastim; Biological: pegfilgrastim; Drug: lyso-thermosensitive liposomal doxorubicin(Thermodox); Procedure: hyperthermia treatment

INTERVENTIONS:
Biological: filgrastim
Biological: pegfilgrastim
Drug: lyso-thermosensitive liposomal doxorubicin(Thermodox)
Procedure: hyperthermia treatment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as liposomal doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Hyperthermia therapy kills tumor cells by heating them to several degrees above normal body temperature. Giving temperature-sensitive liposomal doxorubicin together with hyperthermia may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of temperature-sensitive liposomal doxorubicin when given together with hyperthermia in treating women with locally recurrent breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of temperature-sensitive liposomal doxorubicin (ThermoDox™) when used in combination with local-regional hyperthermia in women with locally recurrent breast cancer.
* Determine the pharmacokinetic profile of ThermoDox™ when used in multiple-course dosing.

OUTLINE: This is a dose-escalation study of temperature-sensitive liposomal doxorubicin (ThermoDox™).

Patients receive ThermoDox™ IV over 30 minutes immediately followed by hyperthermia to the chest wall/axilla over 1-2 hours on day 1. Treatment repeats every 21-35 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of ThermoDox™ (with or without standard-dose granulocyte colony-stimulating factor [G-CSF] support) until the maximum tolerated dose (MTD) is determined. The MTD without G-CSF support is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT). At least 6 patients are treated at the MTD. If the only DLT is neutropenia in > 1 of 6 patients treated at any dose level, then additional cohorts of 3-6 patients receive escalating doses of ThermoDox™ with G-CSF support (standard-dose G-CSF or standard-dose pegfilgrastim) until the MTD is determined. The MTD with G-CSF support is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience DLT after the addition of G-CSF support.

Quality of life and pain are assessed at baseline, prior to courses 3 and 5, and at 21-42 days after completion of therapy.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Locally recurrent disease involving the chest wall and/or its overlying skin

    * Clinically and biopsy proven disease on the chest wall area measuring ≥ 1 cm
    * Overall surface extent of tumor ≤ two 16 x 16 cm fields
    * Tumor thickness ≤ 3 cm by clinical exam and CT scan or MRI
    * Disease extent on the chest wall that exceeds the above criteria allowed provided no other local therapies are available
    * Patients with axillary disease involvement only must meet the above criteria in order to be eligible
    * Prior skin changes consistent with inflammatory breast cancer are allowed
* Distant metastasis (excluding known brain metastases) allowed

  * No resectable chest wall recurrence as the only site of metastatic disease
  * No refractory pain secondary to metastatic disease
* Must have undergone prior local radiotherapy to the chest wall or breast in the adjuvant or metastatic setting
* Must have progressed on ≥ 1 course of hormonal therapy for metastatic disease (if tumor is estrogen receptor positive or progesterone receptor positive) AND ≥ 1 course of chemotherapy
* Prior contralateral breast malignancy allowed provided not previously treated with chemotherapy
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Zubrod performance status 0-1 OR Karnofsky performance status 90-100%
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Bilirubin normal
* alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* left ventricular ejection fraction (LVEF) ≥ 50% by multiple gated acquisition scan (MUGA) or echocardiogram
* No nonhealing wounds or active infection in the area of the chest wall
* No clinically significant findings on baseline evaluations, including laboratory and physical examinations, vital signs, and ECG
* No prior sensitivity (e.g., rash, dyspnea, wheezing, urticaria, or other symptoms) attributed to anthracyclines or other liposomally encapsulated drugs
* No other prior or concurrent primary malignancy except for melanoma in situ, nonmelanoma skin cancer, squamous cell carcinoma, or noninvasive cervical carcinoma
* No history of any of the following:

  * Cardiac ischemia or acute coronary artery syndrome, myocardial infarction (MI), cerebral vascular accident, or abnormal cardiac stress testing within the last 6 months
  * Coronary artery disease (including non-Q wave MI)
  * Uncontrolled hypertension or cardiomyopathy
  * Cardiac valvular surgery or open heart surgery
  * Known structural heart disease
* No other serious medical illness including, but not limited to, the following:

  * Congestive heart failure
  * Life-threatening cardiac arrhythmias
  * Acute or chronic liver disease
* No major psychiatric illness that required inpatient treatment within the past 3 months or that would preclude obtaining informed consent
* No concurrent devices or conditions that might interfere with the hyperthermia portion of the trial, including any of the following:

  * Functioning cardiac pacemaker
  * Metal plates, rods, or prosthesis of the chest wall
  * Severe numbness and/or tingling of the chest wall or breast
  * Skin grafts and/or flaps on the breast or chest wall
  * Unstable cardiovascular or pulmonary status
* No known allergy to eggs or egg products

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 months since prior major surgery
* No prior therapy with anthracyclines exceeding the following doses:

  * Doxorubicin hydrochloride > 450 mg/m^2
  * Epirubicin hydrochloride > 900 mg/m^2
* More than 42 days since prior trastuzumab (Herceptin®)
* More than 90 days since prior radiotherapy to the involved chest wall area
* No other concurrent systemic anticancer therapy, including hormonal therapy, chemotherapy, or investigational anticancer therapy
* No concurrent radiotherapy, including radiotherapy for pain control
* No concurrent administration of any of the following drugs:

  * Amphotericin B by injection
  * Antithyroid agents
  * Azathioprine
  * Chloramphenicol
  * Colchicine
  * Flucytosine
  * Ganciclovir
  * Interferon
  * Plicamycin
  * Zidovudine
  * Sulfinpyrazone
  * Probenecid
  * Cyclosporine
  * Phenobarbital
  * Phenytoin
  * Streptozocin
  * Live vaccines
* Concurrent bisphosphonates for palliation of bony metastasis allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of temperature-sensitive liposomal doxorubicin (ThermoDox™) in combination with hyperthermia | 4 years

SECONDARY OUTCOMES:
Pharmacokinetics | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly L. Blackwell, MD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

REFERENCES:
- [Result] Nolen BM, Marks JR, Ta'san S, Rand A, Luong TM, Wang Y, Blackwell K, Lokshin AE. Serum biomarker profiles and response to neoadjuvant chemotherapy for locally advanced breast cancer. Breast Cancer Res. 2008;10(3):R45. doi: 10.1186/bcr2096. Epub 2008 May 12. PMID 18474099
- [Derived] Zagar TM, Vujaskovic Z, Formenti S, Rugo H, Muggia F, O'Connor B, Myerson R, Stauffer P, Hsu IC, Diederich C, Straube W, Boss MK, Boico A, Craciunescu O, Maccarini P, Needham D, Borys N, Blackwell KL, Dewhirst MW. Two phase I dose-escalation/pharmacokinetics studies of low temperature liposomal doxorubicin (LTLD) and mild local hyperthermia in heavily pretreated patients with local regionally recurrent breast cancer. Int J Hyperthermia. 2014 Aug;30(5):285-94. doi: 10.3109/02656736.2014.936049. PMID 25144817